CLINICAL TRIAL: NCT02210143
Title: An Explorative Study To Develop A Predictive Model Based On Avascular Exposed Root Surface Area For Root Coverage
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Prof., Cukurova University
Other Study IDs: CUDHF-2011-8-6
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (3):
- AERSA-I gingival recession: The AERSA classification was developed based on 15 mm2 which is the lowest cut-off point and the group of AERSA ≤ 15 mm2 named as AERSA-I (low risk group)
- AERSA-II gingival recession: AERSA > 15 mm2 named as AERSA-II (high risk group).
- Miller gingival recession: Gingival recessions classified according to Miller

SUMMARY:
The aim of this study was to evaluate the reliability of the avascular root surface area as a prognostic identification criterion for gingival recessions and to compare the predictive value of the Miller classification and avascular root surface area (AERSA) calculation on the final root coverage outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of isolated Miller I, II or III recession, (Miller 1985a)
* Presence of identifiable cementoenamel junction (CEJ); presence of a step ≤ 2mm at CEJ level and/or the presence of a root abrasion, but with an identifiable CEJ,
* Full-mouth plaque score and Full-mouth bleeding score of < 15% (four sites/tooth),
* No occlusal interferences;
* Non-smokers

Exclusion Criteria:

* Tooth with a prosthetic restoration involving CEJ,
* Patients with a history of periodontitis or abscess formation,
* Presence of systemic disease or taking medications known to interfere with periodontal tissue health
* Pregnant or nursing patients

Ages: 21 Years to 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Ninety one patients, 41 females and 50 males, aged between 21-41 years, with 91 isolated single gingival recessions (32 Miller I, 29 Miller II, 30 Miller III defects) located at upper and lower incisors and canines.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months

SECONDARY OUTCOMES:
mean root coverage | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University Ethics Comitee, Adana, Balcali, Turkey (Türkiye)